CLINICAL TRIAL: NCT03996239
Title: Exercise as Interception Therapy: A "Proof-of-Concept" Digitized Trail
Brief Title: Researching the Effect of Aerobic Exercise on Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-126
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Cancer
Keywords: Aerobic Exercise; 19-126
MeSH Terms: conditions — Neoplasms | interventions — Exercise; Walking; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: For cohort 3 only. Men with histologically-confirmed localized prostate cancer undergoing active surveillance. Both patients and investigators will be fully blinded to the ctDNA status of patients during study participation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- patients with clonal hematopoiesis (Experimental): Exercise treatment will consist of individualized walking delivered up to 5 times weekly. Patients in all cohorts will receive one dose of exercise (i.e., ~300 mins/wk following a non-linear dosing schedule) in both cohorts. Patients will have the option to receive exercise treatment at MSK or at their residence. Home-based exercise will be implemented and monitored using a telemedicine approach (i.e.,TeleEx) established in the Exercise-Oncology (ExOnc) Service
  Interventions: Behavioral: exercise (walking); Other: blood draw
- post treatment patients with breast or colorectal cancer (Experimental): Exercise treatment will consist of individualized walking delivered up to 5 times weekly. Patients in all cohorts will receive one dose of exercise (i.e., ~300 mins/wk following a non-linear dosing schedule) in both cohorts. Patients will have the option to receive exercise treatment at MSK or at their residence. Home-based exercise will be implemented and monitored using a telemedicine approach (i.e.,TeleEx) established in the Exercise-Oncology (ExOnc) Service
  Interventions: Behavioral: exercise (walking); Other: plasma samples; Other: blood draw
- men with localized prostate cancer undergoing active surveillance (Experimental): Exercise treatment will consist of individualized walking delivered up to 5 times weekly. Patients in all cohorts will receive one dose of exercise (i.e., ~300 mins/wk following a non-linear dosing schedule) in both cohorts. Patients will have the option to receive exercise treatment at MSK or at their residence. Home-based exercise will be implemented and monitored using a telemedicine approach (i.e.,TeleEx) established in the Exercise-Oncology (ExOnc) Service
  Interventions: Behavioral: exercise (walking); Other: plasma samples; Other: blood draw
- Individuals with Lynch Syndrome (Experimental): Exercise treatment will consist of individualized walking delivered up to 5 times weekly. Patients in all cohorts will receive one dose of exercise (i.e., ~300 mins/wk following a non-linear dosing schedule) in both cohorts. Patients will have the option to receive exercise treatment at MSK or at their residence. Home-based exercise will be implemented and monitored using a telemedicine approach (i.e.,TeleEx) established in the Exercise-Oncology (ExOnc) Service
  Interventions: Behavioral: exercise (walking); Other: plasma samples; Other: blood draw
- Individuals enrolled on Early Drug Development (EDD) trials (Experimental): Participants will receive structured exercise therapy for 24 weeks. Participants will be followed by standard of care clinical follow-up
  Interventions: Behavioral: exercise (walking)

INTERVENTIONS:
Behavioral: exercise (walking) — Exercise treatment will consist of individualized walking delivered up to 5 times weekly. This trial will evaluate one dose of exercise (i.e., ~300 mins/wk following a non-linear dosing schedule) in both cohorts. Patients will have the option to receive exercise treatment at MSK or at their residence. Home-based exercise will be implemented and monitored using a telemedicine approach (i.e.,TeleEx) established in the Exercise-Oncology (ExOnc) Service
Other: plasma samples — Plasma samples will be obtained at baseline.
  Arms: Individuals with Lynch Syndrome; men with localized prostate cancer undergoing active surveillance; post treatment patients with breast or colorectal cancer
Other: blood draw — fasting blood
  Arms: Individuals with Lynch Syndrome; men with localized prostate cancer undergoing active surveillance; patients with clonal hematopoiesis; post treatment patients with breast or colorectal cancer

SUMMARY:
This study is being done to answer the following question: Will aerobic exercise (exercise that stimulates and strengthens the heart and lungs, and improves the body's use of oxygen) change the biomarkers (signs of disease) found in the blood?

ELIGIBILITY:
Inclusion Criteria:

Cohort 1: CH

* CH called by MSK practices as documented by an MSK physician
* Age ≥18 yrs
* Completion of all anticancer therapy
* High risk of cardiovascular disease defined by presence of at least one of the following:

  * Age ≥60
  * Prior treatment with chemotherapy
  * Prior left-sided breast and/or chest wall radiotherapy
  * Currently receiving or previously received androgen deprivation therapy Prior bone marrow transplant
  * History of smoking
  * Currently treated for one or more cardiovascular risk factors (i.e., hypertension, diabetes, hyperlipidemia)
* Performing less than 150 minutes of structured moderate-intensity or strenuous-intensity exercise per week, as evaluated by self-report
* Willingness to comply with all study-related procedures

Cohort 2: Solid Tumor

* Patients at risk of harboring circulating tumor DNA as defined by one of the following:

  * Histologically confirmed stage III (i.e., high risk of recurrence) colorectal cancer within 2 years of completion of all adjuvant therapy.
  * Histologically confirmed stage III breast cancer with residual disease after neoadjuvant therapy and within 12 months of completing (neo)adjuvant chemotherapy
  * Patients with metastatic breast cancer and radiographic stable disease or NED for ≥6 months and not currently receiving chemotherapy (endocrine therapy and anti-HER2 antibodies allowed)
* Age ≥ 18 yrs
* Performing less than 150 minutes of structured moderate-intensity or strenuous-intensity exercise per week, as evaluated by self-report
* Willingness to comply with all study-related procedures

Cohort 3: Active Surveillance

* Men with histologically confirmed localized prostate cancer undergoing active surveillance
* Age ≥ 18 yrs
* Performing less than 15 minutes of structured moderate-intensity or strenuous-intensity exercise per week, as evaluated by self-report
* Willingness to comply with all study-related procedures
* Cleared for exercise participation as per pre-screening clearance via PAR-Q+

Cohort 4: Lynch Syndrome

* Age ≥18 yrs
* Hereditary colorectal cancer syndrome, specifically Lynch syndrome, defined by the presence of a deleterious germline mutation in the MLH1, MSH2, MSH6, PMS2 or EPCAM genes
* Have a portion of the distal colon or rectosigmoid intact to enable collection of normal mucosa biopsies
* Performing less than 150 minutes of structured moderate-intensity or strenuous-intensity exercise per week, as evaluated by self-report
* Willingness to comply with all study-related procedures
* Cleared for exercise participation as per pre-screening clearance via PAR-Q+

Cohort 5: EDD Phase 0a

* Age ≥18 yrs
* Receiving investigational agent under an EDD protocol for at least 2 months.
* Performing less than 150 minutes of structured moderate-intensity or strenuous-intensity exercise per week, as evaluated by self-report
* Willingness to comply with all study-related procedures
* Cleared for exercise participation as per pre-screening clearance via PAR-Q+

Phase 0b

* Age ≥18 yrs
* Newly Within 3 months of initiating investigational agent on an EDD Service protocol
* Performing less than 150 minutes of structured moderate-intensity or strenuous-intensity exercise per week, as evaluated by self-report
* Willingness to comply with all study-related procedures
* Cleared for exercise participation as per pre-screening clearance via PAR-Q+

Exclusion Criteria:

* Concurrent use of any form of antitumor therapy (endocrine therapy and anti-HER2 antibodies allowed)
* Enrollment onto any other interventional investigational study except interventions determined by the PI not to confound study outcomes (does not apply to Cohort 5: EDD)
* Any other condition or intercurrent illness that, in the opinion of the investigator, makes the subject a poor candidate for study participation.
* Mental impairment leading to inability to cooperate
* Any of the following contraindications to cardiopulmonary exercise testing (Cohorts 1 and 2 only):

  1. Acute myocardial infarction within 3-5 days of any planned study procedures;
  2. Unstable angina
  3. Uncontrolled arrhythmia causing symptoms or hemodynamic compromise
  4. Recurrent syncope
  5. Active endocarditis
  6. Acute myocarditis or pericarditis
  7. Symptomatic severe aortic stenosis
  8. Uncontrolled heart failure
  9. Acute pulmonary embolus or pulmonary infarction within 3 months of any planned study procedures
  10. Thrombosis of lower extremities within 3 months of any planned study procedures
  11. Suspected dissecting aneurysm
  12. Uncontrolled asthma
  13. Pulmonary edema
  14. Respiratory failure
  15. Acute non-cardiopulmonary disorders that may affect exercise performance
* Room air desaturation at rest ≤ 85% (Cohorts 1 and 2 only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
number of patients with variant allele frequency (VAF) | 2 years
  measured by targeted CH panel in peripheral blood
changes in residual tumor burden (Solid tumor group) | 2 years
  measured by the amount of circulating tumor DNA (ctDNA)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - University of California, Los Angeles (Data or Specimen Analysis Only), Los Angeles, California
  - SOMALOGIC (Data or Specimen Analysis Only), Boulder, Colorado
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - LABORATORY CORPORATION OF AMERICA HOLDINGS (Data or Specimen Analysis Only), Burlington, North Carolina
  - Duke University Medical Center (Data or Specimen Analysis Only), Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm